CLINICAL TRIAL: NCT01129167
Title: Frequency of Methods of Local Invasion of Pancreatic Adenocarcinoma
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Other Study IDs: AAAD6885
Record Dates: First submitted 2010-05-21; First posted 2010-05-24 (Estimated); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic adenocarcinoma; Local invasion by pancreatic adenocarcinoma; Recurrence of pancreatic cancer; Surgical resection of pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pancreatic cancer often spreads through local invasion into local structures, including fat, blood vessels, nerves, and nearby organs (stomach, duodenum, spleen, bile duct). Local microscopic invasion is associated with recurrence of pancreatic cancer after pancreatic resection, such that even if the original cancer is surgically removed, microscopic areas of cancer often remain. Data on the patterns of local invasion by pancreatic cancer have not been published. In this study, The investigators hope to investigate the frequency of the various methods of local invasion of pancreatic adenocarcinoma. This would help the investigators better understand how pancreatic cancer spreads, and determine what cancers are not resectable.

DETAILED DESCRIPTION:
Pancreatic cancer is the eighth most common malignancy, and the fifth leading cause of cancer-related death, in the United States. Unfortunately, patients often present late in the course of the disease. Accordingly, the 1- year survival rate is approximately 20%, and the 5-year survival rate is less than 4%. Even in patients with local disease who are surgical candidates, survival at five years remains only 10-25%. Staging for pancreatic adenocarcinoma typically utilizes the TNM classification, where "T" represents tumor size, "N" represents regional lymph node metastasis, and "M" represents distant metastasis. This type of staging can usually only be done after operative resection. Unfortunately, up to 25% of patients are found to be unresectable at the time of surgical exploration. This is most often due to local invasion or metastatic disease. Local microscopic invasion is associated with recurrence of pancreatic cancer after pancreatic resection. Comprehensive data on the patterns of local invasion by pancreatic cancer have not been published. The investigators believe that it would be beneficial to investigate the frequency of the various methods of local invasion of pancreatic adenocarcinoma. A clearer understanding of the natural history of local invasion could potentially lead to a better determination of what constitutes unresectability.

ELIGIBILITY:
Inclusion Criteria:

* Tissue confirmed diagnosis of pancreatic adenocarcinoma.
* Underwent surgical resection for adenocarcinoma at the Columbia University Medical Center between 2001-2009.

Exclusion Criteria:

* Did not undergo surgery.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population will include patients who have been diagnosed with pancreatic adenocarcinoma and who are undergoing surgical resection at CUMC.
Sampling Method: Non-Probability Sample
Enrollment: 1052 (Actual)
Dates: Start 2009-09-15 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Frequency of local invasion modalities in surgical population | 1 year
  The clinical and pathology information from the CUMC surgical database will be reviewed to determine the frequency of the various modalities of local invasion of pancreatic adenocarcinoma. This includes: peripancreatic fat invasion, neural/perineural invasion, vascular invasion, macrovascular invasion, duodenal invasion, bile duct invasion, splenic invasion,and gastric invasion.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy K Chung, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No